CLINICAL TRIAL: NCT03285139
Title: Peer Administered Group Cognitive Behavioural Therapy for Postpartum Depression
Brief Title: Peer Administered CBT for PPD
Acronym: PL-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Kids Can Fly Brantford (Unknown)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, Assistant Professor, Department of Psychiatry and Behavioural Neurosciences, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PL CBT
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Postpartum Depression
Keywords: Postpartum depression; CBT; Lay Peer
MeSH Terms: conditions — Depression, Postpartum | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate Intervention (Experimental): Group CBT for PPD. Women in the treatment group will attend a 9-week group Cognitive Behavioural Therapy intervention for PPD. This intervention was developed at the Women's Health Concerns Clinic (WHCC) at St. Joseph's Healthcare Hamilton and designed to be brief, simple, and applicable to women in community settings. It consists of 9 weekly 2-hour sessions where core CBT skills are learned and practiced, and a new psychoeducational topic is introduced and discussed by women each week. The CBT intervention will be delivered by lay-peers.
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Wait List Controls (Experimental): Group CBT for PPD 9 weeks after enrollment. The women in this arm of the study will receive the same Cognitive Behavioural Therapy intervention as in the immediate intervention arm, however they will begin the CBT group 9 weeks after enrolling in the study.
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Healthy Controls (No Intervention): No treatment. The participants in this arm of the study will not be suffering from postpartum depression and will not receive the Cognitive Behavioural Therapy treatment. Healthy controls will complete study measures upon enrollment in the study, 9 weeks later as well as 6 months later.

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — Cognitive Behavioral Therapy 9 weekly 2-hour group CBT sessions delivered by trained lay peers.
  Arms: Immediate Intervention; Wait List Controls

SUMMARY:
Postpartum depression (PPD) affects up to 20% of women and has profound effects on mothers and their infants. Unfortunately, fewer than 15% of women with PPD receive evidence-based care. This is at least partly due to significant difficulties faced by women in accessing cognitive behavioural therapy (CBT), a preferred 1st line treatment. In Ontario at present, there is a significant lack of personnel trained to deliver CBT. This study will utilize a randomized controlled trial design (with wait list controls) and recruit 70 participants to determine if women with a past history of PPD (i.e., lay peers) can be trained to deliver effective group CBT to women with current PPD. If peers can be trained to provide effective CBT, more women would receive treatment and the burden of PPD on women, families, and the healthcare system would be significantly reduced.

DETAILED DESCRIPTION:
Postpartum depression (PPD) affects up to 20% of women and has profound effects on mothers and their infants. Indeed, the cost of one case of PPD is estimated to exceed $150,000. Unfortunately, fewer than 15% of women with PPD receive evidence-based care and this is at least partly due to difficulties accessing treatment, particularly those that are most preferred (e.g., psychotherapy).

Clinical practice guidelines recommend that the majority of women with PPD receive psychotherapy (e.g., cognitive behavioural therapy (CBT)) as a 1st-line treatment and that screening only occur in settings where CBT is readily available. In order to increase access to treatment, screening efforts have been undertaken by public health units province-wide. This is despite recommendations that this only be conducted in the setting of timely access to evidence-based psychotherapies (e.g., CBT). The purpose of this study is to apply task shifting to the treatment of PPD by determining if women with a past history of PPD (i.e., lay peers) living in the community can be trained to deliver effective group CBT to women with current PPD.

A group CBT intervention for PPD has been developed and validated as well as a training program that pilot data suggests is capable of successfully training public health nurses with little background psychiatric training. This intervention is brief, effective, and generalizable to women with PPD in community. Peer administered interventions (PAIs), those delivered by recovered former patients are increasingly recognized as potentially effective alternatives to traditional mental health care services. Eight lay peers will be trained to deliver our 9-week group CBT treatment. 74 women will be recruited and using a randomized controlled trial design (with wait list controls), it will be determined if lay peers can deliver effective group CBT for PPD.

If peers can be trained to provide effective CBT, more women would receive treatment and the burden of PPD on women, families, and the healthcare system would be significantly reduced. Providing women with PPD with CBT skills at this crucial stage in life also has the capacity to prevent future depressive relapse with significant benefits for patients, families, employers, and the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Eligible women will be >18 years of age, understand and speak English (so that they can participate in the CBT group and complete study measures), have an EPDS score between 10 and 23. They will also all be within 12 months of delivering an infant.

Exclusion Criteria:

* Women can have psychiatric commodities with the exception of bipolar disorder, a current psychotic, substance or alcohol use disorder, or antisocial or borderline personality disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | 6 months
  The EPDS will be used to assess maternal depression. A score of >12 is consistent with PPD and changes in scores >4 are indicative of clinically significant improvement.

SECONDARY OUTCOMES:
Postpartum Bonding Questionnaire | 6 months
  Used to detect disorders of the mother-infant relationship.
Social Provisions Scale | 6 months
  Used to measure the degree to which mothers' social relationships provide support.
CCHS Maternal Healthcare Utilization | 6 months
  Adopted from the Canadian Community Health Survey to Track use of healthcare services by mothers and their infant.
Adult Adolescent Parenting Inventory | 6 months
  Used to assess the parenting and child rearing attitudes of parents.
Cognitive Therapy Awareness Scale | 6 months
  Used to assess CBT skill and knowledge and fidelity to the CBT model.
Therapist Evaluation Checklist | 6 months
  Used to assess the quality of CBT practice.
EQ-5D | 6 months
  Used to measure health-related quality of life.
Generalized Anxiety Disorder-7 | 6 months
  Used to assess generalized anxiety disorder, the most common comorbidity of postpartum depression.
Mini International Neuropsychiatric Interview - Current Major Depressive Disorder | 6 months
  Used to asses maternal depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Van Lieshout, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Kids Can Fly, Brantford, Ontario, Canada

REFERENCES:
- [Derived] Amani B, Merza D, Savoy C, Streiner D, Bieling P, Ferro MA, Van Lieshout RJ. Peer-Delivered Cognitive-Behavioral Therapy for Postpartum Depression: A Randomized Controlled Trial. J Clin Psychiatry. 2021 Nov 9;83(1):21m13928. doi: 10.4088/JCP.21m13928. PMID 34758210